CLINICAL TRIAL: NCT03048747
Title: A Multicenter, Uncontrolled, Open-label, Dose-titration Trial to Investigate the Efficacy and Safety of Tolvaptan Tablets in Patients With Hyponatremia in Syndrome of Inappropriate Antidiuretic Hormone Secretion (SIADH)
Brief Title: A Multicenter Trial to Investigate the Efficacy and Safety of Tolvaptan in Patients With Hyponatremia in SIADH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-14-003; JapicCTI-173512 (Other: Japic)
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Syndrome of Inappropriate Antidiuretic Hormone Secretion
MeSH Terms: conditions — Inappropriate ADH Syndrome | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tolvaptan (Experimental): Tolvaptan tablets at 7.5, 15, 30 (one tablet each), or 60 mg (two 30 mg tablets) will be orally administered once daily after breakfast for up to 30 days.
  Interventions: Drug: Tolvaptan Oral Tablet

INTERVENTIONS:
Drug: Tolvaptan Oral Tablet — Tolvaptan tablets at 7.5, 15, 30 (one tablet each), or 60 mg (two 30 mg tablets) will be orally administered once daily after breakfast for up to 30 days.

SUMMARY:
The objective of this study is to investigate the efficacy and safety of tolvaptan based on the change in serum sodium concentration following administration of tolvaptan oral tablets at 7.5 to 60 mg/day for up to 30 days in patients with hyponatremia in the SIADH.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a definite diagnosis of SIADH in reference to "Diagnostic and Treatment Manual of the Hypersecretion of Vasopressin (SIADH), Revised in 2011"
* Subjects who have been on fluid restriction for at least 7 consecutive days at the time of informed consent and who are showing no improvement of hyponatremia at the time of the screening examination

Exclusion Criteria:

* Subjects who have transient hyponatremia induced by drug administration
* Subjects who are unable to sense thirst or who have difficulty with fluid intake
* Subjects with urinary tract obstruction
* Subjects who have participated in any other clinical trial within 30 days prior to informed consent
* Subjects with serum sodium concentration of <120 mEq/L associated with neurologic impairment, including apathy, confusion, or seizures

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Japan (6):
  - Chubu Region
  - Chugoku Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Sikoku Region

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
  Supporting Materials: Study Protocol and Statistical Analysis Plan (SAP) Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
  Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available aftermarketing approval in global markets, or beginning1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and Ranalytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 16 participants from 31 trial sites in Japan.
Pre-assignment Details: Adults with a definite diagnosis of SIADH in reference to "Diagnostic and Treatment Manual of the Hypersecretion of Vasopressin (SIADH), Revised in 2011"
Period: Overall Study
Arm/Group | Tolvaptan
Started | 16
Completed | 11
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Participant Met Withdrawal Criteria | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set, which included in patients who received ≥1 dose of the study medication.
Arm/Group | Tolvaptan
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 16
Region of Enrollment [Number; unit: participants]
  Japan | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Normalized Serum Sodium Concentration on the Day After Final IMP Administration
Description: The percentage of subjects with normalized serum sodium concentration, defined as ≥135 mEq/L, on the day after final IMP administration will be calculated versus the number of subjects with serum sodium concentration of <135 mEq/L at baseline on Day 1 of the treatment period.
Time Frame: Baseline, Day2, Day3, Day4, Day5, Day7, Day14, Day21, Day after final study medication
Population: Efficacy sample consisted of all participants who received at least one dose of study medication and have Baseline and at least one Post-Baseline efficacy evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 16
percentage of participants
  Day2 | 43.8
  Day3: number analyzed (Participants) | 15
  Day3 | 80
  Day4: number analyzed (Participants) | 15
  Day4 | 80
  Day5: number analyzed (Participants) | 14
  Day5 | 85.7
  Day7: number analyzed (Participants) | 14
  Day7 | 92.9
  Day14: number analyzed (Participants) | 12
  Day14 | 83.3
  Day21: number analyzed (Participants) | 11
  Day21 | 81.8
  Day after final study medication | 81.3

2. Secondary Outcome: Change in Serum Sodium Concentration
Description: The mean and standard error of measured values for serum sodium concentration on the day of fixing the maintenance dose and on the day after final IMP administration were calculated.
  The day of fixing the maintenance dose: Day2, Day3, Day4, Day5, Day7, Day14, and Day21
Time Frame: Day2, Day3, Day4, Day5, Day7, Day14, Day21 and the day after final IMP administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mEq/L
Groups:
- Tolvaptan: Tolvaptan
Arm/Group | Tolvaptan
Number analyzed (Participants) | 16
mEq/L
  Day2 | 6.9 (2.6)
  Day3: number analyzed (Participants) | 15
  Day3 | 8.1 (3.8)
  Day4: number analyzed (Participants) | 15
  Day4 | 8.5 (4.6)
  Day5: number analyzed (Participants) | 14
  Day5 | 8.8 (4.4)
  Day7: number analyzed (Participants) | 14
  Day7 | 10.0 (4.5)
  Day14: number analyzed (Participants) | 12
  Day14 | 10.8 (3.7)
  Day21: number analyzed (Participants) | 12
  Day21 | 10.4 (6.0)
  Day after final study medication | 11.0 (4.3)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from signing of the informed consent form until follow-up, up to 7 weeks on average.
Description: A serious adverse event (SAE) was an untoward medical occurrence that resulted in death or required inpatient hospitalization or prolonged hospitalization. An AE was an exacerbation of an existing problem or a new problem experienced by a participant when enrolled in a trial whether or not it was considered drug related by study physician.
Arm/Group | Tolvaptan
All-Cause Mortality (participants affected / at risk) | 1/16
Serious Adverse Events (participants affected / at risk) | 5/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (N=16)
Supraventricular extrasystoles (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Bacteraemia (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Loss of consciousness (Nervous system disorders) | 1
Paralysis of recurrent laryngeal nerve (Nervous system disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (N=16)
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Cerumen impaction (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Anorectal disorder (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Malaise (General disorders) | 1
Pyrexia (General disorders) | 2
Thirst (General disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 1
Bacteaemia (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 2
Periodontitis (Infections and infestations) | 1
Skin bacterial Infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Blood alanine phoshatase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood sodium increased (Investigations) | 1
Nuetrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Weight decreased (Investigations) | 2
White blood cell count increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
hypocalcaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Headache (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Paralysis recurrent Laryngeal nerve (Nervous system disorders) | 1
Depressive symptom (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Bladder disoder (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rapid correction of hyponatremia (Surgical and medical procedures) | 1
Circulatory collapse (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT03048747/SAP_000.pdf
  • Study Protocol (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT03048747/Prot_001.pdf